CLINICAL TRIAL: NCT03163342
Title: Extent and Durability of Immune Response Following Seasonal Influenza Vaccination in Healthy Volunteers
Brief Title: Immune Response Following Seasonal Influenza Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Collaborators: Optimal Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALT-FLZ-401
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Influenza
Keywords: Seasonal
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open label (Other): Licensed seasonal influenza vaccine, intramuscular
  Interventions: Biological: Licensed seasonal influenza vaccine

INTERVENTIONS:
Biological: Licensed seasonal influenza vaccine — 20 healthy subjects will be enrolled and receive a single dose of licensed seasonal influenza vaccine

SUMMARY:
This is an open-label, single administration dose study in adult healthy male and female subjects. After qualifying for the study, subjects will receive a single intramuscular injection of the FDA approved 2016-2017 quadrivalent influenza vaccine.

DETAILED DESCRIPTION:
Subjects will be screened within 28 days prior to enrollment into the study. After qualifying for the study subjects will visit the clinical unit on Day l and will have pre-dose blood samples taken for humoral (serum) and cellular(peripheral blood mononuclear cells PBMCs) immunity testing and nasopharyngeal swabs for assessment of mucosa! immunity, and will then be given the vaccine.

Over the next 6 months, I 0-mL blood samples will be collected on Days 4, 8, 15, 29, 91 and 181 for HAI testing. Peripheral blood mononuclear cells will be collected on Day 8 to assess cellular responses. A nasopharyngeal swab will also be done on Day 29. Screening assessments will include clinical laboratory tests (hematology, chemistry, urinalysis (UA), drug and alcohol testing), vital signs, 12-lead electrocardiogram and physical examination.

Adverse events (AEs) will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 to 50 years of age, inclusive
2. Good general health status, as determined by the Investigator
3. Adequate venous access for repeated phlebotomies
4. Screening laboratory results within institutional normal range or Grade 1 elevation if the Investigator documents clinical insignificance. Bilirubin may be Grade 2 if associated with no1mal alanine aminotransferase (ALT) and aspartate aminotransferase (AST) and the Investigator considers the result not to be clinically significant (e.g. vigorous exercise or Gilbert's syndrome)
5. Negative drug and alcohol screen at Screening and pre-dose on Day I
6. For women of child bearing potential, negative pregnancy test
7. Willingness to practice a highly effective method of contraception that may include, but is not limited to, abstinence, sex only with persons of the same sex,monogamous relationship with a postmenopausal partner, monogamous relationship with vasectomized partner, vasectomy, surgical sterilization (hysterectomy, or bilateral tubal ligation, salpingectomy, or oophorectomy), licensed hormonal methods, intrauterine device (IUD), or consistent use of a barrier method (e.g., condom, diaphragm) with spermicide for 28 days after the Fluzone Intramuscular Quadrivalent vaccine dose.

Exclusion Criteria:

1. Pregnant, possibly pregnant, or lactating women
2. Body mass index> 35.0 kg/m2
3. Positive results for HIV, hepatitis B vims, or hepatitis C virus at Screening
4. Asthma or other chronic lung disease that is greater than mild in severity. Specifically excluded are participants with any of the following events in the past year:

   * Daily symptoms
   * Daily use of short acting beta 2 agonists
   * Use of inhaled steroids or theophylline
   * Use of pulse systemic steroids
   * Emergency care or hospitalization related to asthma or other chronic lung disease
   * Systemic steroids for asthma exacerbation
5. History of diabetes mellitus (gestational diabetes is allowed if treatment was not required postpartum and serum glucose is currently in the normal range)
6. History of coronary artery disease, arrhythmia, or congestive heart failure
7. Clinically significant ECG abnormality
8. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 95 mmHg) at Screening or pre-dose on Day I
9. History of anaphylaxis or angioedema
10. Known allergy to any of the ingredients in the vaccine formulation including egg allergy
11. History of chronic rhinitis, nasal septal defect,cleft palate, nasal polyps, or other nasal abnormality that might affect vaccine administration
12. Previous nasal surgery or nasal cauterization
13. Any symptoms of upper respiratory infection or temperature> 38°C within 3 days before Day I
14. Significant nasal congestion or rhinorrhea as assessed by the investigator.
15. Known or suspected malignancy, excluding non-melanoma skin cancers and other early stage surgically excised malignancies that the Investigator considers to be exceedingly unlikely to recur
16. Immunocompromised individuals, including those who have used corticosteroids (including intranasal steroids), alkylating drugs, antimetabolites, radiation, immune-modulating biologics, or other immunomodulating therapies within 90 days before Day 1 or those who plan use during the study period
17. Use of statin medication within 30 days before Day I (including atorvastatin, fluvastatin,lovastatin, pravastatin, rosuvastatin, simvastatin, pitavastatin)
18. Receipt of intranasal medications (including over-the-counter medications) within 30 days before Day 1
19. Receipt of any IP within 30 days before Day 1
20. Receipt of any vaccine within 30 days before Day I
21. Receipt of intranasal vaccine within 90 days before Day I
22. Receipt of any influenza vaccine within 6 months before Day I
23. Any change in medication for a chronic medical condition within 30 days before Day I
24. Past regular use or current use of intranasal illicit drugs or any regular use of illicit drugs by any other route.
25. Use of tobacco products or electronic cigarettes within 30 days before Day l. Any other smoking products including marijuana will be excluded.
26. Any medical, psychiatric, or social condition or any occupational or other responsibility that in the judgment of the Investigator would interfere with or serve as a contraindication to protocol adherence, assessment of safety (including immunogenicity), or a subject's ability to give informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Bart, MD, Principal Investigator — Optimal Health Research
Locations (1):
- Optimal Health Research, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 34.2 [21 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: HAI Antibody Immune Response to Matched Influenza Strain H1N1 A/California/04/2009 Strain
Description: To evaluate antibody response against matched influenza strain H1N1 A/California/04/2009 strain as measured by hemagglutination inhibition (HAI) following administration of a seasonal influenza vaccine.
Time Frame: Day 29 after vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Groups:
- FluZone: Open label
Arm/Group | FluZone
Number analyzed (Participants) | 20
Geometric Mean Titer | 293.4 [186.7 to 461.3]

2. Secondary Outcome: Antibody Response to Divergent Influenza Strains
Description: l) antibody responses to divergent influenza strains as measured by hemagglutination inhibition (HAI) following administration of a seasonal influenza vaccine
Time Frame: Day 29 after vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | FluZone
Number analyzed (Participants) | 20
GMT
  A/Brisbane/59/2007 (H1 strain) | 12.3 [6.9 to 21.8]
  A/New Jersey/76 (H1 strain) | 37.3 [22.5 to 61.9]
  A/Saint-Petersburg/61/2015 (H1 strain) | 40.7 [21.8 to 76.1]
  A/Vietnam/1203/2004XPR8 (H5 strain) | 9.3 [6.0 to 14.6]

3. Secondary Outcome: Cellular Immune Response
Description: To evaluate cellular immune responses to influenza as measured by PBMC ELISpot following administration of seasonal influenza vaccine
Time Frame: Day 8 after vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | FluZone
Number analyzed (Participants) | 20
GMT | 37.1 [14.3 to 96.2]

4. Secondary Outcome: Mucosal Influenza Antibody Response
Description: To evaluate mucosal influenza antibody responses as measured by IgA ELISA following administration of seasonal influenza vaccine
Time Frame: Day 29 after vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | FluZone
Number analyzed (Participants) | 20
GMT | 1.8 [1.2 to 2.7]

ADVERSE EVENTS:
Time Frame: Day 1 through Day 181
Arm/Group | FluZone
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT03163342/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT03163342/SAP_001.pdf